CLINICAL TRIAL: NCT04346290
Title: Effects of Dexmedetomidine on Microcirculation and Residual Kidney Function in Kidney Donors and Transplanted Kidney Function in Kidney Recipients
Brief Title: Effects of Dexmedetomidine on Microcirculation and Residual Kidney Function in Kidney Donors
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201912073MINB
Record Dates: First submitted 2020-03-02; First posted 2020-04-15 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Kidney Transplant; Microcirculation
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standard anesthesia care for kidney donor
- Dexmedetomidine (Experimental): Standard anesthesia care and perioperative infusion of dexmedetomidine for kidney donor
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Initial infusion dose of dexmedetomidine is 0.4 mcg/kg/min, maintenance infusion dose is 0.1-0.7 mcg/kg/min
  Arms: Dexmedetomidine

SUMMARY:
Kidney transplant can help patients with end-stage kidney disease to get rid of dialysis and have a good quality life. However, during the renal donation operation, the stress response and subsequent inflammatory responses may result in damage to the residual kidney and transplanted kidney. Dexmedetomidine can increase urine output and decrease the neutrophil gelatinase associated lipocalin level in patients receiving coronary artery bypass surgery. The primary goal of this trial is to investigate the effects of perioperative infusion of dexmedetomidine on the microcirculation and residual kidney function in kidney donors and on the transplanted kidney function in kidney recipients.

DETAILED DESCRIPTION:
Kidney transplant can help patients with end-stage kidney disease to get rid of dialysis and have a good quality life. However, during the renal donation operation, the stress response and subsequent inflammatory responses may result in damage to the residual kidney and transplanted kidney. In addition, the transplanted kidney will encounter ischemic and reperfusion injuries during kidney transplant, and it may affect its function. It has been reported in several animal studies that dexmedetomidine can reduce microcirculatory dysfunction, kidney injury, and intestinal injury. Moreover, dexmedetomidine can increase urine output and decrease the neutrophil gelatinase associated lipocalin level in patients receiving coronary artery bypass surgery. The primary goal of this trial is to investigate the effects of perioperative infusion of dexmedetomidine on the microcirculation and residual kidney function in kidney donors and on the transplanted kidney function in kidney recipients. This is a single blind and randomized controlled trial. The participants will be randomly assigned to the Control group or Dexmedetomidine group. The participants in the Control group will receive standard anesthesia care for kidney donation operation. Beside the standard anesthesia care, the participants in the Dexmedetomidine group will receive continuously intravascular infusion of dexmedetomidine since 10 minutes after anesthesia till one hour after operation. At several specific time points, participants will receive sublingual microcirculation examination by using an incident dark field video microscope and blood tests. The chart information will be recorded. The blood creatinine level of the kidney donors and recipients at 1 and 6 months will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Kidney Donor for living kidney transplant

Exclusion Criteria:

* Allergy to dexmedetomidine
* Severe bradycardia < 50 beats per minute before surgery
* Severe atrioventricular block (the second or third degree)
* Non-native speaker

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-07-24 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Change of perfused vessel density | Postoperative 1 hour
  Sublingual microcirculation is measured by incidental dark field video microscope (CytoCam). Perfused vessel density is equal to perfused vessel length (in millimeter) divided by total vessel length (in millimeter) in a square millimeter.

SECONDARY OUTCOMES:
Change of creatinine level | Postoperative 1 day
  change of creatinine level between preoperative and postoperative level
Change of perfused vessel density | Postoperative 1 day
  Sublingual microcirculation is measured by incidental dark field video microscope (CytoCam). Perfused vessel density is equal to perfused vessel length (in millimeter) divided by total vessel length (in millimeter) in a square millimeter.
Change of creatinine level | Postoperative 1 month
  change of creatinine level between preoperative and postoperative level
Change of creatinine level | Postoperative 6 months
  change of creatinine level between preoperative and postoperative level

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chang Yeh, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data that underlie results in a publication could be requested.
Supporting Information: Study Protocol, CSR
Time Frame: Starting 6 months after publication for two years
Access Criteria: Principal investigator will review requests. The criteria for reviewing requests includes research purpose and methods of data protection.